CLINICAL TRIAL: NCT05683119
Title: The Effect of Menstrual Cycle and Oral Contraceptive Pill Phase on Aspects of Exercise Physiology and Athletic Performance in Female Athletes
Brief Title: The Effect of Menstrual Cycle and Oral Contraceptive Pill Phase on Aspects of Exercise Physiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 120869
Record Dates: First submitted 2022-10-20; First posted 2023-01-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Menstrual Cycle; Oral Contraceptives
Keywords: Athletic performance; Exercise physiology; Female; Athlete
MeSH Terms: interventions — Exercise; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This study will conduct the same outcome measures in two populations (i.e., eumenorrheic women and OCP users).
Who Masked: Outcomes Assessor
Masking Description: The experimenter will be blind to the intended testing timepoint. Experimenter blinding will be achieved by having an independent party schedule the testing session, based on the participant's hormonal profile, without disclosing this to the experimenter who will conduct the testing session. On completion of the study, the blinded experimenters will be asked to comment if blinding was achieved and maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUM Group (Experimental): Participants must: have menstrual cycle lengths ≥ 21 days and ≤ 35 days resulting in 9 or more consecutive periods per year; provide evidence of a luteinising hormone (LH) surge; demonstrate the required hormonal profile as defined below; and have not used any type of hormonal contraceptives (HC) for a minimum of 3 months, but ideally 6 months, prior to enrolment.
  Phase 1- Indicated by the onset of bleeding until day 5 Oestrogen and progesterone levels are low
  Phase 2- Oestrogen higher than during phase 1 and 3 Progesterone higher than during phase 1, but lower than 6.36 nmol·L-1 Must be followed by a positive luteinising hormone surge
  Phase 3- +7 days after ovulation has been confirmed Oestrogen higher than phase 1, but lower than phase 2 Progesterone >16 nmol·L-1
  Interventions: Other: Exercise and blood draw
- OCP Group (Experimental): Participants must: have been taking their OCP ≥ 3 months prior to recruitment; be taking a combined, monophasic, second generation OCP; and demonstrate the correct hormonal profile as defined below.
  Pill-taking phase- Indicated by the 21 consecutive pill-taking days Oestrogen and progesterone levels are low; ≤ phase 1 of the menstrual cycle
  Pill-free phase- Indicated by the 7 consecutive pill-free days Oestrogen and progesterone levels may begin to rise in comparison with the pill-taking phase
  Interventions: Other: Exercise and blood draw

INTERVENTIONS:
Other: Exercise and blood draw — This project intends to investigate the effects of circulating fluctuations in oestradiol and progesterone, experienced during the menstrual cycle [MC] and oral contraceptive pill [OCP] use, on aspects of exercise physiology and athletic performance in female athletes. This research aims to determine if a particular hormonal profile affects physiological functioning (e.g., muscle strength, maximum oxygen uptake) and/or athletic performance in female athletes. The intervention will include a stretching regimen, balance test, push-ups, agility test, handgrip muscle test, vertical jump, flexibility test, cycling protocol, blood sample and height/ weight measurements.

SUMMARY:
This study will investigate the effect of menstrual cycle (MC) and oral contraceptive pill phase on aspects of exercise physiology and athletic performance in female athletes. Specifically, this study intends to investigate the effects of circulating fluctuations in oestradiol and progesterone, experienced during the menstrual cycle and oral contraceptive pill use, on aspects of exercise physiology and athletic performance in female athletes. This research will help researchers determine if a particular hormonal profile affects physiological functioning such as muscle strength, maximum oxygen uptake and athletic performance in female athletes.

DETAILED DESCRIPTION:
The menstrual cycle is the body's way of preparing for pregnancy. A "normal" or "healthy" cycle lasts an average of 21-35 days, which starts on the first day of bleeding. Throughout each cycle, levels of the hormones oestrogen and progesterone vary. The oral contraceptive pill is designed to prevent pregnancy; one way it does this is by lowering the levels of oestrogen and progesterone. The main purpose of oestrogen and progesterone is for reproduction. These hormones have also been shown to affect other bodily functions. The effects of oestrogen and progesterone on a woman's capacity to undertake exercise is an important factor for active women to consider to optimise training schedules and athletic performances. Emerging research has suggested that menstrual cycle phase or oral contraceptive use is associated with changes in sport and exercise performance. However, research on this topic is lacking (both in quality and quantity), and currently is quite contradictory. Much more high-quality research is required to explore the impact of both natural and supplemented oestrogen and progesterone on exercise-related outcomes to give convincing advice to active women. This research must follow strict procedural guidelines and include accurate hormonal measurement (through blood samples) to increase its usefulness to exercising women. Such research is needed to establish a cause-and-effect relationship for any differences in exercise physiology and athletic performance between the different phases of the menstrual cycle, between phases of oral contraceptive pill taking and not-taking, and between women using or not-using oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Cis gender women
* 18-40 years of age
* Body mass index ≥ 19.5 and ≤ 25 kg∙-2; an exception can be made in the case of some athletes where they have a higher BMI, but are considered more lean/muscular than fat.
* Must be defined as healthy, i.e., not having any medical condition or taking any medication known to affect any of the outcome measures. Examples include diagnosed hyperandrogenism from polycystic ovary syndrome, congenital adrenal hyperplasia, or other differences in sexual development.
* Cannot smoke
* Considered to be physically active. Participants training status will be classified using the criteria outlined by McKay et al. (In press). For this study, participants must be Tier 2 athletes or above (Table 1). In addition, participants will be considered on the basis of relative maximal oxygen consumption (Decroix et al., 2016); needing to be Performance Level 2 or above (Table 2). Participants must provide details on gravidity and parity and must not be in the postpartum period (i.e., within 12 months of childbirth), currently breastfeeding, or pregnant. Participants will be recruited based on their endogenous hormonal profile (i.e., eumenorrheic or OCP users) and these profiles (including inclusion/exclusion criteria) are described below in detail.

Group Specific Inclusion Criteria:

Group 1. Eumenorrheic [EUM]

* Must have menstrual cycle lengths ≥ 21 days and ≤ 35 days resulting in 9 or more consecutive periods per year
* Must provide evidence of a luteinising hormone (LH) surge
* Must demonstrate the required hormonal profile as defined in Table 3
* Cannot have used any type of hormonal contraceptives (HC) for a minimum of 3 months, but ideally 6 months, prior to enrolment

Group 2. Oral contraceptive pill [OCP] users

* Must have been taking their OCP ≥ 3 months prior to recruitment
* Must be taking a combined, monophasic, second generation OCP (see Table 4 for permitted brands)
* Must demonstrate the correct hormonal profile as defined in Table 5

Exclusion Criteria:

-Cannot speak, read and understand English

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood Sample | Every visit (9-10 blood draws depending on the group). Through study completion, an average of 5 months.
  A blood sample will be drawn by a trained phlebotomist from an antecubital vein. Approximately 10 mL will be collected.
Cycling Protocol | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  Prior to and following the cycling protocol a note will be made of any unique details of the test environment (i.e., temperature, humidity, pressure), performance, or athlete concerns in the comments section of the data sheet. Participants will complete a 5-minute warm-up at 35 W.
  Phase 1:
  The protocol will commence at a power output of 45 W and increased by 15 W every 4 min. For each stage, power output, average heart rate (HR) in the last 30 seconds, and blood lactate values in the last 15 seconds will be recorded. The last completed 4-minute workload will be recorded as maximal 4-minute power output.
  Phase 2:
Height | First visit only- Month 1
  Height will be measured in bare feet, with minimal clothing, and no impeding hairstyles, using a stadiometer. Participants will be positioned in the 'Frankfort Plane' and will be asked to take a deep breath, which they hold, while the measurement is taken.
Weight | Through study completion, an average of 5 months.
  Body mass will be measured at every testing session by an experimenter using the same scales on each occasion (i.e., within and between participants) and the participants wearing minimal clothing and no shoes.
Stork Balance Stand Test | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  Participants are required to remove their shoes and place their hands on their hips, then position their non-supporting foot against the inside knee of the supporting leg. They will be given one minute to practice the balance. Participants must raise their heel to balance on the ball of their foot. The stopwatch is started as the heel is raised from the floor. The stopwatch is stopped if any of the follow occur:
  * the hand(s) come off the hips
  * the supporting foot swivels or moves (hops) in any direction
  * the non-supporting foot loses contact with the knee
  * the heel of the supporting foot touches the floor The total time in seconds is recorded. The score is the best of three attempts. Allow 1 minute rest between attempts. Participants may continue to perform the test (beyond three attempts) as long as improvements are being made.
Muscular Endurance: Push-ups | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  The push-up test is administered with participants starting in a modified knee push-up position (legs together, lower leg in contact with the mat and ankles plantar flexed, back straight, hands shoulder width apart, head up, using the knees as the pivotal point). The participants must raise the body by straightening the elbows and return to the "down" position, until the chin touches the mat. The stomach should not touch the mat. The participant's back must be straight at all times and the participant must push up to a straight arm position. The maximum number of push-ups performed consecutively without rest is counted as the score. The test is stopped when the participant strains forcibly or unable to maintain the appropriate technique within two repetitions.
Illinois Agility Test | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  The length of the course is 10 meters and the width is 5 meters. Four cones are used to mark the start, finish and the two turning points. Another four cones are placed down the centre an equal distance apart. Each cone in the centre is spaced 3.3 meters apart. You will be asked to lie on your front (head to the start line) with your hands by your shoulders. On the 'Go' command the stopwatch is started, and you must get up as quickly as possible and run around the course in the direction indicated, without knocking the cones over, to the finish line, at which the timing is stopped. The total time in seconds is recorded. The score is the best of three attempts. Allow 1 minute rest between attempts. Participants may continue to perform the test (beyond three attempts) as long as improvements are being made.
Muscular Strength: Handgrip | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  The participant holds the dynamometer in the dominant hand, with the arm at right angles and the elbow by the side of the body. The handle of the dynamometer is adjusted if required - the base should rest on the first metacarpal (heel of palm), while the handle should rest on middle of the four fingers. When ready the participant squeezes the dynamometer with maximum isometric effort, which is maintained for about 5 seconds. No other body movement is allowed. The participant should be strongly encouraged to give a maximum effort. The score is the best of three attempts. Allow 1 minute rest between attempts. Participants may continue to perform the test (beyond three attempts) as long as improvements are being made.
Countermovement (power) jump | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  This test will be administered using the My Jump 2 app, which calculates the height, flight time, velocity, force, and power of vertical jumps by recording the jump and selecting accurately its take-off and landing. All participants will follow the same jump protocol. The participant squats down until the knees are bent at 90 degrees, then immediately jumps vertically as high as possible, landing back on the mat on both feet at the same time. Allow one minute rest between trials. The take-off must be from both feet, with no initial steps or shuffling. The best result of three attempts is recorded - participants may continue to jump (beyond three attempts) as long as improvements are being made. It is also important that the athlete not only jumps as high as possible, but also attempts to land in the same position as they took off - as jumping forwards, backwards or sideways can affect the test results.
Sit and Reach Flexibility Test | Visits 2-9 (EUM Group) and Visits 3, 5, 7-10 (OCP Group). Through study completion, an average of 5 months.
  This test involves sitting on the floor with legs stretched out straight ahead. Shoes should be removed. The soles of the feet are placed flat against the box. Both knees should be locked and pressed flat to the floor - the tester may assist by holding them down. With the palms facing downwards, and the hands on top of each other or side by side, you must reach forward along the measuring line as far as possible. Ensure that the hands remain at the same level, not one reaching further forward than the other. After some practice reaches, you must reach out and hold that position for one-two seconds while the distance is recorded. Make sure there are no jerky movements. The score is the best of three attempts. Allow 1 minute rest between attempts. Participants may continue to perform the test (beyond three attempts) as long as improvements are being made.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Thornton, Principal Investigator — Schulich-Family Medicine
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No